CLINICAL TRIAL: NCT05117814
Title: Zanubrutinib Monotherapy in Relapsed/Refractory Central Nervous System Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Associate Chief of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-2001-IIT
Record Dates: First submitted 2021-09-25; First posted 2021-11-11 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: CNS Lymphoma
Keywords: CNSL
MeSH Terms: interventions — zanubrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrtuinib (Experimental): Zanubrutinib 320mg Qd
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — as long as 24 months or consolidated with ASCT or WBRT after achieving PR or CR
  Other Names: BGB-3111; BRUKINSA®

SUMMARY:
Zanubrutinib is a novel BTK inhibitor with proven activity in patients with various B-cell lymphomas addicted to the B-cell receptor signaling pathway.

DETAILED DESCRIPTION:
Studies involving gene expression profiling and next generation sequencing have demonstrated that CNS lymphomas mostly are of the ABC-subtype and harbor mutations that reinforce BCR signaling. Ibrutinib, as the first BTK inhibitor, showed substantial activity in patients with R/R PCNSL and R/R SCNSL. Zanubrutinib is a novel BTK inhibitor with proven activity in patients with various B-cell lymphomas addicted to the B-cell receptor signaling pathway. In addition, pharmacological studies demonstrated the free drug exposure of zanubrutinib at 160 mg BID is roughly 10 times that of ibrutinib at 560 mg QD, and penetration into the CNS by zanubrutinib and ibrutinib is similar, suggesting the potential activity of zanubrutinib in the treatment of CNS lymphomas. However, the outcome of R/R PCNSL and R/R SCNSL patients treated with zanubrutinib monotherapy is still unclear.

ELIGIBILITY:
Inclusion Criteria:

Key inclusion criteria:

1. Able to understand and willing to sign a written informed consent document
2. Men and woman at least 18 years of age on the day of consenting to the study
3. Histologically documented DLBCL.
4. Relapsed/refractory PCNSL or relapsed/refractory SCNSL
5. Patients with parenchymal lesions must have unequivocal evidence of disease progression on imaging (MRI or the brain or head CT) prior to study enrollment. For patients with leptomeningeal disease only, CSF cytology must document lymphoma cells and/or imaging findings consistent with CSF disease prior to study enrollment.
6. An ECOG performance status≤2
7. Adequate bone marrow and organ function shown by:

(1) Neutrophils ≥ 0.75 x 109/L independent of growth factor support within 7 days of study entry (2) Platelets ≥ 50 x 109/L independent of growth factor support or transfusion within 7 days of study entry (3) Creatinine clearance of ≥ 30 mL/min (4) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN) (5) Bilirubin ≤ 1.5 x ULN (6) International normalized ratio ≤ 1.5 and activated partial thromboplastin time ≤ 1.5 x ULN.

8. Recovered to grade 1 toxicity from prior therapy before the first dose of study drug 9. Agree to use highly effective methods of birth control during the period of therapy and for 3 months after the last dose of the study drug.

Exclusion Criteria:

1. Patients with SCNSL actively receiving treatment for extra-CNS disease
2. Concurrently using other approved or investigational antineoplastic agents
3. Prior chemotherapy, targeted therapy, or radiation therapy within 4 weeks
4. Prior exposure to a BTK inhibitor
5. Concurrently using more than 8mg of dexamethasone daily or the equivalent
6. History of other active malignancies within 2 years of study entry
7. Major surgery within 4 weeks of screening or not recovered from the side effects of such surgery
8. Known to have human immunodeficiency virus (HIV) infection
9. Known to have a history of active or chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) as determined by serologic tests
10. Active infection systemic including infections requiring oral or intravenous antimicrobials
11. Currently active clinically significant cardiovascular disease
12. QTcF > 480 msecs or other significant electrocardiogram (ECG) abnormalities
13. Unable to swallow capsules or disease significantly affecting gastrointestinal function
14. Any life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could have compromised the patient's safety, or put the study at risk
15. Required ongoing treatment with medication that are strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitors or strong CYP3A inducers
16. History of stroke or intracranial hemorrhage within 6 months prior to enrollment
17. Inability to comply with study procedures
18. Pregnant or lactating women
19. Prior allogenic hematopoietic stem cell transplantation (autologous stem cell transplant is NOT an exclusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 2 years
  Based on the Investigator assessed CR and PR, with the enhanced CT scan, the cerebrospinal fluid (CSF) examination, and the ophthalmological examination.

SECONDARY OUTCOMES:
Time to response (TTR) | 2 years
  Time from the first dose of zanubrutinib to the first assessment of >=PR
Duration of response (DOR) | 2 years
  Time from the first assessment of >=PR to symptom, CT scan, and/ or CSF confirmed progressive disease (PD)
The concentration of zanunbrutinib in CSF and plasma | 2 months
  The concentration of zanunbrutinib in CSF and plasma 2 hours after taking the drug
Progression-free survival (PFS) | 2 years
  The time from the first dose to PD or death whichever occurs earlier.
Treatment-related adverse events (TRAE) | During zanubrutinib treatment until 30+/-7 days after discontinuation.
  Adverse events during zanubrutinib treatment.

OTHER OUTCOMES:
Overall survival (OS) | 4 years
  The time from the first dose to death.
ctDNA | 2 years
  ctDNA In CSF.

CONTACTS AND LOCATIONS:
Overall Officials: Shenmiao Yang, MD, Principal Investigator — Peking University Peoples' Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China